CLINICAL TRIAL: NCT03965663
Title: Vibro-tactile Pressure Feedback of the Prosthetic Foot for Trans-tibial Amputees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Agnes Sturma (Other)
Collaborators: University of Applied Sciences Upper Austria (Other)
Responsible Party: Sponsor-Investigator, Agnes Sturma, Physical Therapist, Research Fellow, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2238/2017
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-tibial Amputees (Experimental): Unilateral Trans-tibial Amputees that use vibro-tactile feedback for six months in daily living
  Interventions: Device: Vibro-tactile Feedback
- Trans-tibial Amputees with TSR (Experimental): Unilateral Trans-tibial Amputees that use vibro-tactile feedback for six months in daily living. The subjects underwent a functional nerv-transfer surgery prior to participation, where the proximal part of the sural nerv was to the distal part of the saphenous nerv.
  Interventions: Device: Vibro-tactile Feedback

INTERVENTIONS:
Device: Vibro-tactile Feedback — The device measures the force between the prosthetic food and the ground. With this signals, vibratators are triggered. The vibrators are housed by the prosthetic socket and stimulate the stump.

SUMMARY:
The aim of the study is to investigate the influence of a vibro-tactile device on trans-tibial amputees in terms of gait, pain and perception of the prosthesis.

DETAILED DESCRIPTION:
The study is divided into three phases. The initial phase lasts 6 to 8 weeks for each subject. For subjects of group 2 the length of the initial phase depends on the progression of the re-innervation. The initial phase ends, when the subject can perceive the tactile stimulate at the re-innervated area of the skin. During the initial phase, all subjects get a new prosthesis. To minimize the adjusting to the new prosthesis only a new socket, which houses the vibro-tactile Feedback system, is fabricated and the old prosthetic food is re-used. After a period of 3 weeks minimum, where the subjects use the new prosthesis, a gait analysis and an assessment of the sensitivity of the skin at the stump are performed.

Subsequently the intervention phase starts and the vibro-tactile feedback system is activated. For a period of 6 months the subjects use the new prostheses with the integrated vibro-tactile feedback system in daily living. After 2 and 4 months, the subjects visit the study site for an assessment of the sensitivity of the skin. After 6 months a second gait analysis and an other assessment of the sensitivity of the skin a the stump are performed. Afterwards the vibro-tactile feedback-system is disabled.

During the observing phase the subjects use the prosthesis with the disabled vibro-tactile feedback system for 4 months.

During all three phases the subjects answer the questionnaires every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* unilateral trans-tibial amputation
* uses a prostheses already for more than 1 year
* sufficient touch sensitivity at the stump
* unimpaired contralateral lower extremity

Exclusion Criteria:

* psychiatric disorder
* cognitive restrictions
* pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Trinity Amputation and Prosthesis Experience Scales-Revised (TAPES-R) | 1 year
  The Trinity Amputation and Prosthesis Experience Scales-Revised (TAPES-R) is a multidimensional instrument designed to examine the psychosocial processes involved in adjusting to amputation and a prosthesis. TAPES consists of 9 subscales, with possible scores depending on the single subscale. The range is from 0-12 to 0-25 (depending on the number of items and answer possibilities).

SECONDARY OUTCOMES:
Fall Efficacy Scale International Version (FES-I) | 1 year
  The Fall Efficacy Scale International Version (FES-I) is a questionaire that assesses the fear of falling. Scores can range from 16-64, with a higher score indicating a higher fear of falling.
Pain Visual analoge scale (VAS) | 1 year
  The pain is measured with a Visual analoge scale form 0 to 10. O indicates no pain, while 10 is the worst pain the person can imagine.
Number of falls within the last two months | 1 Year
  Subjects report the number a falls within the last two months.
Gait parameters | 6 months
  Two gait analysis are performed with a 3D video-based marker system. Standard gait parameters (as cardence, speed, step length and weight) as well as kinematic and kinetic parameters are calculated.
two point discrimination | 6 months
  the two point discrimination (in mm) at the skin of the stump is assessed
touch perception threshold | 6 months
  the touch percertion at the skin of the stump is assessed with mono filaments

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Sturma, MSc, Study Director — Medical University Vienna

IPD SHARING:
Plan to Share IPD: Yes
All IPD from the mentioned outcome parameters are planned to be made available to other researchers.
Time Frame: upon publication in a scientific journal